CLINICAL TRIAL: NCT06760351
Title: Bridging Traditional Chinese and Western Medicine: Efficacy, Safety, and Diagnostic Advances in a Pilot Cohort-Based Observational Study for Moderate to Severe Anemia
Brief Title: Pulse Diagnosis and Anemia: Exploring Integrated Traditional Chinese and Western Medicine Approaches
Status: Completed | Type: Observational
Sponsor: Chia-Ying Chuang (Other)
Responsible Party: Sponsor-Investigator, Chia-Ying Chuang, Doctor of Chinese medicine department, Principal Investigator, Resident physician, Taichung Tzu Chi Hospital
Organization: Taichung Tzu Chi Hospital (Other)
Other Study IDs: REC109-61
Record Dates: First submitted 2024-12-29; First posted 2025-01-06 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Moderate to Severe Anemia; Traditional Chinese Medicine (TCM); Pulse Diagnosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Traditional Chinese Medicine (TCM) Group: Participants in this group received individualized TCM herbal formulations tailored to address systemic imbalances observed in moderate to severe anemia. Commonly used formulations include Yougui Wan, Zuogui Wan, and Xiong Gui Jiao Ai Tang. Treatment was monitored monthly with adjustments made based on clinical symptoms and pulse diagnosis parameters.
  Interventions: Drug: TCM Herbal Therapy
- Western Medicine Group: Participants in this group were treated using standard Western medical protocols for moderate to severe anemia. Treatments included blood transfusions and erythropoiesis-stimulating agents when necessary, based on clinical evaluations.
  Interventions: Drug: Standard Western Medicine Treatment

INTERVENTIONS:
Drug: TCM Herbal Therapy — Administration of customized herbal formulations for the TCM group, targeting qi and blood regulation. Pulse diagnosis parameters were evaluated monthly to guide treatment adjustments.
  Groups: Traditional Chinese Medicine (TCM) Group
Drug: Standard Western Medicine Treatment — Administration of standard Western medical care, including blood transfusions and erythropoiesis-stimulating agents, focusing on hemoglobin restoration and anemia management.
  Groups: Western Medicine Group

SUMMARY:
This observational study evaluates the efficacy and safety of integrated Traditional Chinese Medicine (TCM) and Western medicine in managing moderate to severe anemia. The study examines hemoglobin (Hb) level improvements and correlations with TCM pulse diagnosis parameters at six diagnostic positions (Right and Left Chung, Guan, and Chi). Conducted at Taichung Tzu Chi Hospital, it aims to explore TCM's role as a complementary approach to anemia care while maintaining a focus on patient safety and integrated diagnostic techniques.

DETAILED DESCRIPTION:
The study included 28 patients with moderate to severe anemia (Hb < 10 g/dL) treated between February 26, 2021, and December 31, 2022. Participants were divided into two groups: those receiving TCM-based interventions (herbal formulations tailored to address systemic imbalances) and those following standard Western medicine protocols. Data collection involved monthly monitoring of Hb levels and pulse diagnosis parameters using the Huang-T1 Sphygmograph, which provided detailed insights into frequency-domain and waveform-derived characteristics.

Primary outcomes included Hb level improvements and safety assessments, while secondary outcomes focused on the correlations between pulse parameters and hematological changes. Results indicated consistent Hb improvements in the TCM group, with notable trends observed in pulse diagnosis correlations. These findings highlight TCM's potential as a diagnostic and therapeutic adjunct in anemia care, emphasizing its role in bridging traditional and modern medical practices.

The study adheres to ethical guidelines, with approval from the Taichung Tzu Chi Hospital Research Ethics Committee (Approval Number: REC109-61). All participants provided written informed consent prior to study inclusion. Future directions include larger-scale studies and randomized controlled trials to further validate findings and expand their clinical applicability.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of moderate to severe anemia (Hb < 10 g/dL).
* Age between 18 and 90 years.
* Willingness to provide informed consent and comply with study procedures.
* Ability to attend monthly follow-up visits and provide clinical data for analysis.

Exclusion Criteria:

* Presence of psychiatric disorders affecting compliance.
* Significant organ diseases, such as chronic obstructive pulmonary disease, advanced liver disease, or heart failure.
* Pregnancy or lactation.
* Concurrent participation in other clinical trials or use of investigational drugs within the past 30 days.
* Non-compliance with follow-up schedules or study protocols.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with moderate to severe anemia receiving treatment at Taichung Tzu Chi Hospital. Study population includes patients managed under TCM and Western medicine frameworks to evaluate integrated care approaches.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Monthly Change in Hemoglobin Levels (g/dL) to Assess Treatment Efficacy | Baseline to 5 months
  Monthly measurement of hemoglobin levels (g/dL) to evaluate improvements in anemia severity from baseline over a 5-month study period.

SECONDARY OUTCOMES:
Correlation Between Pulse Diagnosis Parameters and Monthly Hemoglobin Levels (g/dL) | Baseline to 5 months
  Analysis of the relationship between pulse parameters (e.g., Right Chi Pulse AIr, Right Chung Pulse D Wave) and Hb levels, using data collected monthly from the Huang-T1 Sphygmograph.
Incidence of Treatment-Related Adverse Events (Safety) | Baseline to 5 months
  Documentation of any adverse events or side effects related to TCM herbal formulations or Western medical treatments, monitored monthly.

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Tzu Chi Hospital, Taichung, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
The following individual participant data (IPD) will be shared: anonymized datasets related to hemoglobin levels, pulse diagnosis parameters, and treatment outcomes. All shared data will be de-identified to ensure participant confidentiality.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: IPD and supporting information will be available starting 6 months after publication of the study results and will remain accessible for 5 years thereafter.
Access Criteria: Researchers with a scientifically valid proposal will be granted access to the IPD and supporting documents. Requests should be submitted to the corresponding author and must include a research plan outlining the intended use of the data. Data will be shared through secure, password-protected platforms.